CLINICAL TRIAL: NCT01363271
Title: Cost Study of Linezolid Versus Vancomycin Among Previously Hospitalized Patients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: University of Maryland (Other); Lodise & Lodise, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: A5951160
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Complicated Skin and Structure Infection; Nosocomial Pneumonia
MeSH Terms: conditions — Healthcare-Associated Pneumonia | interventions — Linezolid; Vancomycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- complicated skin and skin structure infections (cSSSI): Identified through a pre-specified list of ICD-9 codes in study protocol.
  Interventions: Drug: Linezolid; Drug: Vancomycin
- Pneumonia: Identified through a pre-specified list of ICD-9 codes in study protocol.
  Interventions: Drug: Linezolid; Drug: Vancomycin

INTERVENTIONS:
Drug: Linezolid — IV and oral forms of linezolid are identified through a pre-specified list of National Drug Codes (NDCs).
  Groups: complicated skin and skin structure infections (cSSSI)
Drug: Vancomycin — IV form of vancomycin is identified through a pre-specified list of National Drug Codes (NDCs).
  Groups: complicated skin and skin structure infections (cSSSI)
Drug: Linezolid — IV and oral forms of linezolid are identified through a pre-specified list of National Drug Codes (NDCs).
  Groups: Pneumonia
Drug: Vancomycin — IV form of vancomycin is identified through a pre-specified list of National Drug Codes (NDCs).
  Groups: Pneumonia

SUMMARY:
This is a retrospective, observational, non-interventional drug study using de-identified data from two administrative claims datasets. The study design and analysis will reflect the perspective of the commercially insured. The objectives of this study are twofold:

1. To compare the rates of re-hospitalization among patients treated with either linezolid orally or IV, or vancomycin IV for complicated skin and skin structure infections (cSSSI) or pneumonia hospitalization.
2. To compare the total direct medical costs of patients treated with linezolid orally or IV, or vancomycin IV for cSSSI or pneumonia hospitalization.

DETAILED DESCRIPTION:
A sampling method is not used in this study since it is a retrospective, non-interventional claims database analysis. Pre-specified inclusion/exclusion criteria and ICD-9, NDC, HCPC codes are applied to identify the study cohorts.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

* Patients with a hospitalization for cSSSI or pneumonia for which the discharge date (i.e. index date) is between January 1, 2007 and September 30, 2009.
* Patient must have a claim for either vancomycin (IV) or linezolid (IV or oral) within 7 days following their cSSSI or pneumonia hospitalization discharge date (i.e. index date). We will exclude patients who initially receive both vancomycin and linezolid on the same day. We will apply an intention-to-treat approach and use the first drug as the index drug, even if the "comparator drug" (e.g. vancomycin for linezolid and vice-versa) is used subsequently on a future date. If there are both oral and IV formulations of the same index drug on the same index date, the patient will be kept and categorized as an IV user. As with all duplicate claims, for two claims that have both oral and IV index drug as well as the same IV and oral costs on the same index date, the claim with the oral drug will be removed, and the patient will be called an IV user.
* 18-64 years of age at index date.
* Continuous eligibility for six months prior to the index hospitalization date. No minimum of post-index continuous enrolment is required to assure that early mortality patients are included (maximum of 180 days after the index vancomycin or linezolid claim).

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

* Patients who were enrolled in Medicare.
* Patients who were over age 65 or younger than 18.
* Patients with fewer than 3 days of oral therapy.
* Patients with index hospitalization of greater than 30 days.
* Patients with osteomyelitis, infective endocarditis, meningitis, joint infections, necrotizing fasciitis, gangrene, prosthetic joint infection, or prosthetic implant/ device infection during index hospitalization.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of patients with a hospitalization for complicated skin and skin structure infections (cSSSI) or pneumonia. We will identify cases from January 1, 2007, to September 30, 2009, with additional 6 months pre-period and up to 6 months of post-index follow-up period.
Sampling Method: Non-Probability Sample
Enrollment: 7260 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Rehospitalization | 42 days
Total reimbursed amount following hospital discharge | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5951160&StudyName=Cost%20Study%20of%20Linezolid%20Versus%20Vancomycin%20Among%20Previously%20Hospitalized%20Patients